CLINICAL TRIAL: NCT04135937
Title: A Personalized mHealth Approach to Smoking Cessation for Veterans Living With HIV (CDA 17-005)
Brief Title: Mobile Evidence-Based Smoking Cessation for Veterans Living With HIV (MESH)
Acronym: MESH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX 19-002; CDA 17-005 (Other Grant/Funding Number: VA ORD HSR&D)
Record Dates: First submitted 2019-10-17; First posted 2019-10-23 (Actual); Results first posted 2022-02-16 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Human Immunodeficiency Virus; Smoking
Keywords: Human Immunodeficiency Virus; Smoking; Veterans
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Smoking | interventions — Bupropion; Varenicline; Cognitive Behavioral Therapy; Nicotine Replacement Therapy; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- MESH (Experimental): Mobile Evidence-Based Smoking Cessation for Veterans Living with HIV is an intervention that is tailored for participants. It can include cognitive behavioral therapy, relapse-prevention text messaging, and/or pharmacotherapy with nicotine replacement therapy, bupropion, or varenicline.
  Interventions: Drug: Bupropion; Drug: Varenicline; Behavioral: Cognitive Behavioral Therapy; Drug: Nicotine Replacement Therapy; Behavioral: Relapse Prevention Text Messaging

INTERVENTIONS:
Drug: Bupropion — Smoking cessation pharmacotherapy prescribed in accordance with package insert.
  Other Names: Wellbutrin, Zyban
Drug: Varenicline — Smoking cessation pharmacotherapy prescribed in accordance with package insert.
  Other Names: Chantix
Behavioral: Cognitive Behavioral Therapy — Behavioral intervention; modules include identifying reasons for quitting, setting a quit date, breathing relaxation technique, identifying smoking triggers, identifying social support, and education about relapse prevention
  Other Names: CBT
Drug: Nicotine Replacement Therapy — Participants may be prescribed single-formulation NRT (i.e., nicotine patch) or dual NRT (patch + rescue method such as nicotine gum, inhaler, or lozenges).
  Other Names: NRT; nicotine patch; nicotine rescue method
Behavioral: Relapse Prevention Text Messaging — Participants will be invited to utilize SmokefreeVET, a mobile text messaging service for military Veterans trying to quit smoking. The 6- to 8-week program provides 24/7 encouragement, advice, and tips to help smokers quit smoking and stay quit.
  Other Names: SmokefreeVET

SUMMARY:
Smoking is a significant cause of damage to health and quality of life specifically for Veterans with human immunodeficiency virus (HIV). Smoking cessation interventions for this population are lacking. The primary aim of this project is to explore smoking cessation treatment preferences among Veteran smokers living with HIV. The study team will refine the design and content of a smoking cessation treatment for Veteran smokers living with HIV. The intervention uses mobile health and telehealth technology to personalize smoking cessation counseling and medications and provide relapse prevention text messaging.

DETAILED DESCRIPTION:
Although smoking is a significant cause of damage to health and quality of life specifically for Veterans with human immunodeficiency virus (HIV), smoking cessation interventions for this population are lacking. The primary aim of this project is to qualitatively explore smoking cessation treatment preferences among Veteran smokers living with HIV. The study team will refine the design and content of an intervention that uses mobile health and telehealth technology to a)individually personalize smoking cessation counseling and pharmacotherapy, and b) provide relapse prevention messaging support. It is a personalized, tailored, multi-component intervention for smoking cessation specifically designed for Veteran smokers living with HIV.

This project is highly significant given that: 1) smoking is prevalent among and particularly harmful for HIV-positive Veterans; 2) there is a dearth of research on smoking cessation for Veterans with HIV; 3) current approaches to smoking cessation in this population are not effective; 4) as the largest US provider of HIV health services, VHA is an ideal setting; and 5) the proposed intervention follows the VA Blueprint for Excellence, which prioritizes mobile health and treatment personalization to increase reach/efficacy.

ELIGIBILITY:
Inclusion Criteria:

* VHA patient
* HIV positive serostatus
* currently smoking 7 cigarettes per week
* willing to complete study procedures. Exclusion criteria are:

Exclusion Criteria:

* current hospitalization
* acute risk for suicide documented in the medical record
* inability to complete study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M. Wilson, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MESH
Started | 12
Completed | 9
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | MESH
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.08 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Participate in the Post-treatment Interview
Description: Study primary outcomes are qualitative in nature. Participants will be asked to participate in a qualitative interview in which they will be interviewed regarding things they would change about the proposed treatment intervention. These results will be used to inform the treatment development for a randomized controlled trial.
Time Frame: Post-treatment follow-up visit (week 5)
Measure: Count of Participants; unit: Participants
Arm/Group | MESH
Number analyzed (Participants) | 12
Participants | 9

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | MESH
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MESH (N=12)
irritability (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT04135937/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT04135937/ICF_001.pdf